CLINICAL TRIAL: NCT02251665
Title: National Cerebral and Cardiovascular Center (NCVC) Stroke Registry
Status: Active, not recruiting | Type: Observational
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Kazunori Toyoda, Director and Chair, Dept. of Stroke and Cerebrovascular Diseases, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: NationalCardioCenter
Record Dates: First submitted 2014-09-23; First posted 2014-09-29 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Acute
Keywords: Acute ischemic stroke; Acute intracerebral hemorrhage; Transient ischemic attack
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute ischemic stroke, acute ICH, TIA: Consecutive patients with acute ischemic stroke, intracerebral hemorrhage, and transient ischemic attack who are emergently managed in the stroke care unit or stroke units in the National Cerebral and Cardiovascular Center
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — a single-center prospective observational study

SUMMARY:
A single-center registry of patients with acute ischemic stroke, intracerebral hemorrhage, and transient ischemic attack (TIA) who are emergently managed in the stroke care unit in the National Cerebral and Cardiovascular Center (NCVC) to determine change in underlying characteristics, stroke features and severity, process for diagnosis and acute treatment, and long-term outcomes of stroke/TIA patients over the years.

DETAILED DESCRIPTION:
This is a single-center registry of consecutive patients with acute ischemic stroke, intracerebral hemorrhage, and transient ischemic attack (TIA) who are emergently managed in the stroke care unit in the National Cerebral and Cardiovascular Center, a flagship stroke center in Japan.

Neurological emergencies other than stroke/TIA and subclinical cerebrobvascular inpatients are also enrolled.

Data are collected and analyzed to determine change in underlying characteristics, stroke features and severity, process for diagnosis and acute treatment, and long-term outcomes of stroke/TIA patients over the years.

The National Cerebral and Cardiovascular Center was founded in 1977 in Suita, Osaka, in order to provide the public with the most advanced treatment for cardiovascular and cerebrovascular diseases and to conduct the highest level of basic as well as applied research on the cardiovascular and cerebrovascular systems.

ELIGIBILITY:
Inclusion Criteria:

1. A patient with acute ischemic stroke, intracerebral hemorrhage, and transient ischemic attack who are emergently managed in the stroke care unit or stroke units in the National Cerebral and Cardiovascular Center (NCVC)
2. Consent to participate in the registration by a patient or relatives obtained using an opt-out approach by the demonstrating contents of the registration on the hospital bulletin board

Exclusion Criteria:

1) Patients considered by the investigator to be unsuitable for participating in this registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients
Sampling Method: Non-Probability Sample
Enrollment: 5374 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The modified Rankin Scale (mRS), a measure of disability | 3 monhts
  mRS scores range from 0 (no symptoms at all) to 6 (death)

SECONDARY OUTCOMES:
Number of participants | at entry
  Also assessing underlying patients' characteristics prior to index stroke/TIA
National Institutes of Health Stroke Scale score | at entry
  Also assessing neurological and cognitive states
Volume of culprit infarcts/hematoma | at entry
  ASPECTS on DWI for ischemia or hematoma volume using the ABC/2 method
The modified Rankin Scale (mRS), a measure of disability | around 3 weeks
  mRS scores range from 0 (no symptoms at all) to 6 (death). Participants will be followed at hospital discharge, an expected average of 3 weeks.
The modified Rankin Scale (mRS), a measure of disability | 1 year
  mRS scores range from 0 (no symptoms at all) to 6 (death)
Events of cardiovascular diseases including stroke/TIA | around 3 weeks
  Participants will be followed at hospital discharge, an expected average of 3 weeks.
Events of cardiovascular diseases including stroke/TIA | 3 months
Events of cardiovascular diseases including stroke/TIA | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Toyoda, MD, PhD, Principal Investigator — Vice Director of the Hospital, National Cerebral and Cardiovascular Center
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Result] Toyoda K, Ninomiya T. Stroke and cerebrovascular diseases in patients with chronic kidney disease. Lancet Neurol. 2014 Aug;13(8):823-33. doi: 10.1016/S1474-4422(14)70026-2. PMID 25030514
- [Result] Osaki M, Miyashita F, Koga M, Fukuda M, Shigehatake Y, Nagatsuka K, Minematsu K, Toyoda K. Simple clinical predictors of stroke outcome based on National Institutes of Health Stroke scale score during 1-h recombinant tissue-type plasminogen activator infusion. Eur J Neurol. 2014 Mar;21(3):411-8. doi: 10.1111/ene.12294. Epub 2013 Nov 7. PMID 24200315
- [Result] Sakamoto Y, Sato S, Kuronuma Y, Nagatsuka K, Minematsu K, Toyoda K. Factors associated with proximal carotid axis occlusion in patients with acute stroke and atrial fibrillation. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):799-804. doi: 10.1016/j.jstrokecerebrovasdis.2013.07.002. Epub 2013 Oct 6. PMID 24103668
- [Result] Sato S, Uehara T, Hayakawa M, Nagatsuka K, Minematsu K, Toyoda K. Intra- and extracranial atherosclerotic disease in acute spontaneous intracerebral hemorrhage. J Neurol Sci. 2013 Sep 15;332(1-2):116-20. doi: 10.1016/j.jns.2013.06.031. Epub 2013 Jul 13. PMID 23859180
- [Result] Kobayashi J, Uehara T, Toyoda K, Endo K, Ohara T, Fujinami J, Nagatsuka K, Minematsu K. Clinical significance of fluid-attenuated inversion recovery vascular hyperintensities in transient ischemic attack. Stroke. 2013 Jun;44(6):1635-40. doi: 10.1161/STROKEAHA.111.000787. Epub 2013 May 7. PMID 23652273
- [Result] Tanaka K, Koga M, Sato K, Suzuki R, Minematsu K, Toyoda K. Three-dimensional analysis of the left atrial appendage for detecting paroxysmal atrial fibrillation in acute ischemic stroke. Int J Stroke. 2014 Dec;9(8):1045-51. doi: 10.1111/ijs.12268. Epub 2014 Mar 13. PMID 24621380
- [Result] Tomii Y, Toyoda K, Suzuki R, Naganuma M, Fujinami J, Yokota C, Minematsu K. Effects of 24-hour blood pressure and heart rate recorded with ambulatory blood pressure monitoring on recovery from acute ischemic stroke. Stroke. 2011 Dec;42(12):3511-7. doi: 10.1161/STROKEAHA.111.628586. Epub 2011 Sep 29. PMID 21960578
- [Result] Koga M, Arihiro S, Miyashita F, Yamamoto H, Yamada N, Nagatsuka K, Minematsu K, Toyoda K. Factors associated with early recanalization failure following intravenous rt-PA therapy for ischemic stroke. Cerebrovasc Dis. 2013;36(4):299-305. doi: 10.1159/000355054. Epub 2013 Oct 16. PMID 24135558
- [Result] Inoue Y, Miyashita F, Koga M, Minematsu K, Toyoda K. Unclear-onset intracerebral hemorrhage: Clinical characteristics, hematoma features, and outcomes. Int J Stroke. 2017 Dec;12(9):961-968. doi: 10.1177/1747493017702664. Epub 2017 Mar 31. PMID 28361615
- [Derived] Koge J, Tanaka K, Yoshimoto T, Shiozawa M, Ohta T, Satow T, Kataoka H, Ihara M, Koga M, Toyoda K. Mechanical Thrombectomy Beyond 2b Reperfusion: Should We Pursue a Higher Reperfusion Grade after Achievement of 2b? Stroke Vasc Interv Neurol. 2022 Jan 12;2(1):e000196. doi: 10.1161/SVIN.121.000196. eCollection 2022 Jan. PMID 41585290
- [Derived] Yamaguchi E, Yoshimoto T, Ogura S, Saito K, Saito S, Hattori Y, Wasida K, Nishimura K, Toyoda K, Koga M, Ihara M. Association of the RNF213 p.R4810K Variant With the Outer Diameter of Cervical Arteries in Patients With Ischemic Stroke. Stroke Vasc Interv Neurol. 2022 Mar 24;2(6):e000298. doi: 10.1161/SVIN.121.000298. eCollection 2022 Nov. PMID 41582976
- [Derived] Inui R, Koge J, Tanaka K, Yoshimoto T, Shiozawa M, Abe S, Ishiyama H, Imamura H, Nakahara J, Kataoka H, Ihara M, Toyoda K, Koga M. Detrimental effect of anemia after mechanical thrombectomy on functional outcome in patients with ischemic stroke. Front Neurol. 2023 Dec 19;14:1299891. doi: 10.3389/fneur.2023.1299891. eCollection 2023. PMID 38187149
- [Derived] Yoshimoto T, Inoue M, Tanaka K, Koge J, Shiozawa M, Kamogawa N, Ishiyama H, Abe S, Imamura H, Kataoka H, Koga M, Ihara M, Toyoda K. Tmax Mismatch Ratio to Identify Intracranial Atherosclerotic Stenosis-Related Large-Vessel Occlusion Before Endovascular Therapy. J Am Heart Assoc. 2023 Jul 18;12(14):e029899. doi: 10.1161/JAHA.123.029899. Epub 2023 Jul 8. PMID 37421278
- [Derived] Okada T, Yoshimoto T, Wada S, Yoshimura S, Chiba T, Egashira S, Kimura S, Shiozawa M, Inoue M, Ihara M, Toyoda K, Takashima H, Koga M. Intravenous Thrombolysis With Alteplase at 0.6 mg/kg in Patients With Ischemic Stroke Taking Direct Oral Anticoagulants. J Am Heart Assoc. 2022 Oct 4;11(19):e025809. doi: 10.1161/JAHA.122.025809. Epub 2022 Sep 21. PMID 36129032
- [Derived] Koge J, Tanaka K, Yoshimoto T, Shiozawa M, Kushi Y, Ohta T, Satow T, Kataoka H, Ihara M, Koga M, Isobe N, Toyoda K. Internal Carotid Artery Tortuosity: Impact on Mechanical Thrombectomy. Stroke. 2022 Aug;53(8):2458-2467. doi: 10.1161/STROKEAHA.121.037904. Epub 2022 Apr 11. PMID 35400203
- [Derived] Inoue M, Yoshimoto T, Tanaka K, Koge J, Shiozawa M, Nishii T, Ohta Y, Fukuda T, Satow T, Kataoka H, Yamagami H, Ihara M, Koga M, Mlynash M, Albers GW, Toyoda K. Mechanical Thrombectomy Up to 24 Hours in Large Vessel Occlusions and Infarct Velocity Assessment. J Am Heart Assoc. 2021 Dec 21;10(24):e022880. doi: 10.1161/JAHA.121.022880. Epub 2021 Dec 10. PMID 34889115
- [Derived] Yoshimoto T, Shiozawa M, Koge J, Inoue M, Koga M, Ihara M, Toyoda K. Evaluation of Workflow Delays in Stroke Reperfusion Therapy: A Comparison between the Year-Long Pre-COVID-19 Period and the with-COVID-19 Period. J Atheroscler Thromb. 2022 Jul 1;29(7):1095-1107. doi: 10.5551/jat.63090. Epub 2021 Aug 13. PMID 34393139
- [Derived] Koge J, Tanaka K, Yoshimoto T, Shiozawa M, Yamagami H, Satow T, Takahashi JC, Ihara M, Koga M, Kira JI, Toyoda K. Early recurrent ischemic events after mechanical thrombectomy: effect of post-treatment intracranial hemorrhage. J Neurol. 2021 Aug;268(8):2810-2820. doi: 10.1007/s00415-021-10449-1. Epub 2021 Feb 16. PMID 33594451
- [Derived] Yoshimoto T, Inoue M, Yamagami H, Fujita K, Tanaka K, Ando D, Sonoda K, Kamogawa N, Koga M, Ihara M, Toyoda K. Use of Diffusion-Weighted Imaging-Alberta Stroke Program Early Computed Tomography Score (DWI-ASPECTS) and Ischemic Core Volume to Determine the Malignant Profile in Acute Stroke. J Am Heart Assoc. 2019 Nov 19;8(22):e012558. doi: 10.1161/JAHA.119.012558. Epub 2019 Nov 8. PMID 31698986
- [Derived] Fujita K, Tanaka K, Yamagami H, Ide T, Ishiyama H, Sonoda K, Satow T, Takahashi JC, Ihara M, Koga M, Yokota T, Toyoda K. Detrimental Effect of Chronic Hypertension on Leptomeningeal Collateral Flow in Acute Ischemic Stroke. Stroke. 2019 Jul;50(7):1751-1757. doi: 10.1161/STROKEAHA.119.025142. Epub 2019 May 16. PMID 31233392
- [Derived] Takasugi J, Yamagami H, Noguchi T, Morita Y, Tanaka T, Okuno Y, Yasuda S, Toyoda K, Gon Y, Todo K, Sakaguchi M, Nagatsuka K. Detection of Left Ventricular Thrombus by Cardiac Magnetic Resonance in Embolic Stroke of Undetermined Source. Stroke. 2017 Sep;48(9):2434-2440. doi: 10.1161/STROKEAHA.117.018263. Epub 2017 Aug 17. PMID 28818863
- [Derived] Hashimoto T, Hayakawa M, Funatsu N, Yamagami H, Satow T, Takahashi JC, Nagatsuka K, Ishibashi-Ueda H, Kira JI, Toyoda K. Histopathologic Analysis of Retrieved Thrombi Associated With Successful Reperfusion After Acute Stroke Thrombectomy. Stroke. 2016 Dec;47(12):3035-3037. doi: 10.1161/STROKEAHA.116.015228. Epub 2016 Oct 25. PMID 27780903
- See also: Official home page of the National Cerebral and Cardiovascular Center — http://www.ncvc.go.jp/english/index.html